CLINICAL TRIAL: NCT06575530
Title: Efficacy and Safety of Remazolam Besylate in Patients Requiring Mechanical Ventilation Admitted to ICU After Non-cardiac Surgery: Protocol for a Randomized, Controlled No-inferiority Trial
Brief Title: Sedation Efficacy and Safety of Remazolam Besylate in Ventilated Surgical Critically Ill Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIT2024-001-002
Record Dates: First submitted 2024-08-11; First posted 2024-08-28 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-02

CONDITIONS: Effect of Drug; Adverse Drug Event; Mechanical Ventilation Complication; Critical Illness; Surgery; Sedation
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Critical Illness | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- remimazolam besylate group (Experimental): Light sedation will started when the patient admitted to ICU after non-cardiac surgery under general anesthesia with remimazolam besylate which will continuously intravenously pumped at a rate of 0.2-1.0mg/kg/h . Depth of sedation will assessed by RASS hourly to ensure a RASS score of 0 to -2. Adjust the dosage of remimazolam (increase or decrease) based on the RASS score. At the same time, use remifentanil (0.1-0.5/kg/min) as a combination analgesic drug to ensure that the CPOT is ≤2 points. When a satisfactory level of RASS score (0 to -2 points) is still not achieved within the upper limit of remimazolam, a remedial sedation will started using propofol. Researchers assess the patient daily during the ICU stay whether to terminate sedative drug, weaning and extubation, and compete the outcomes assessment.
  Interventions: Drug: Remimazolam Besylate
- Dexmedetomidine hydrochloride group (Active Comparator): Light sedation will started when the patient admitted to ICU after non-cardiac surgery under general anaesthesia with dexmedetomidine, which will continuously intravenously pumped at a rate of 0.2-0.7ug/kg/h. Depth of sedation will assessed by RASS hourly to ensure a RASS score of 0 to -2. Adjust the dosage of dexmedetomidine (increase or decrease) based on the RASS score. At the same time, use remifentanil (0.1-0.5/kg/min) as a combination analgesic drug to ensure that the CPOT is ≤2 points. When a satisfactory level of RASS score (0 to -2 points) is still not achieved within upper limit of dexmedetomidine, a remedial sedation will started using propofol. Researchers assess the patient daily during the ICU stay whether to terminate sedative drug, weaning and extubation, and compete the outcomes assessment.
  Interventions: Drug: Dexmedetomidine Hydrochloride

INTERVENTIONS:
Drug: Remimazolam Besylate — patients will be sedated with remimazolam via intravenous pump on the day of ICU admission, the dosage will titrate with the depth of sedation evaluated with RASS. A remedial sedation protocol will be initiated if remimazolam fails to achieve a satisfactory RASS score (0 to -2 points) within its upper dosage limits, propofol will be administered intravenously at a dose of 0.2 mg, followed by reassessment 5 minutes post-injection. The same dose of propofol will be repeated if the desired sedation depth is not reached. Continuous infusion of propofol will be started at a rate of 0.2 to 1 mg/kg/h if satisfactory sedation is not attained after three consecutive intravenous injections of propofol, the continuous infusion will be discontinued once the RASS score reaching the acceptable range (0 to -2).
  Arms: remimazolam besylate group
Drug: Dexmedetomidine Hydrochloride — patients will be sedated with dexmedetomidine hydrochloride via intravenous pump on the day of ICU admission, the dosage will titrate with the depth of sedation evaluated with RASS. A remedial sedation protocol will be initiated if dexmedetomidine fails to achieve a satisfactory RASS score (0 to -2 points) within the upper dosage limits, propofol will be administered intravenously at a dose of 0.2 mg, followed by reassessment 5 minutes post-injection. The same dose of propofol will be repeated if the desired sedation depth is not reached. Continuous infusion of propofol will be started at a rate of 0.2 to 1 mg/kg/h if satisfactory sedation is not attained after three consecutive intravenous injections of propofol, the continuous infusion will be discontinued once the RASS score reaching the acceptable range (0 to -2).
  Arms: Dexmedetomidine hydrochloride group

SUMMARY:
A multi-center, prospective, randomized, double-blind, no-inferiority clinical trial designed to assess the the safety and efficacy of remazolam besylate in sedation of critically ill mechanically ventilated patients after surgery compared to dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old
* must accept no-cardiac elective surgery
* must under general anaesthesia
* can be combined regional tissue anesthesia
* must admitted to ICU with tracheal intubation after general anaesthesia - expected mechanical ventilation time must more than 24 hours
* light or moderate sedation must needed

Exclusion Criteria:

* intracranial surgery or severe neurological or spinal cord disease
* schizophrenia, epilepsy, and Parkinson's disease
* coma, severe dementia, or language barrier before surgery
* cardiac dysfunction or arrhythmia
* severe liver dysfunction(Child-Pugh C class)
* severe kidney dysfunction
* use of dexmedetomidine or remifentanil besylate 24 hours before or during surgery
* pregnancy or lactation
* any investigational drug useage 30 days before surgery
* refuse to participant.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 306 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
ventilation free days | Through the initiation of enrollment to 28 days, an average of 1 day
  ventilation free days(VFDs) at 28 days. VFDs=0 if subject dies within 28 days of mechaincal ventilation; VFDs=28-X if successfully liberated from ventilation X days after initiation; VFDs=0 if the subject is mechaincally ventilated for >28 days.

SECONDARY OUTCOMES:
Dosage of remedial sedatives | Through the useage of sedative drugs in the ICU, an average of 3 days
  Dosage of remedial sedatives during mechanical ventilation in the ICU
Frequency of remedial sedatives | Through the useage of sedative drugs in the ICU, an average of 3 days
  Frequency of remedial sedatives during mechanical ventilation in the ICU
Delirium incidence | Through the ICU stay, an average of 3 days
  Delirium incidence during the patients' ICU stay, assessed using ConfusionAssessmentMethodfortheIntensive CareUnit(CAM-ICU, 4 items), delirium is diagnosed when 3 items are met
Proportional of predicted sedation time | Through the useage of sedative drugs in the ICU, an average of 3 days
  Proportional of predicted sedation time during sedation time in the ICU, sedation depth is assessed using Richmond Agitation Sedation Scale(RASS, -5 to +4), predicted sedation must has a RASS score -2 to 0.
Extubation time after termination of sedation | From ICU admission to extubation, an average of 3 days
  Extubation time(hour) after termination of sedation
Re-mechanical ventilation incidence after weaning and extubation | Through the ICU stay, an average of 3 days
  Re-mechanical ventilation incidence after weaning and extubation
Proportion of different oxygen therapies after extubation | Through the ICU stay, an average of 3 days
  Proportion of different oxygen therapies after extubation
Pain assessment score the first 3 days after surgery | The first 3 days of ICU stay, an average of 3 days
  Pain assessment score the first 3 days after surgery, assessed using Critical-Care Pain Observation Tool(CPOT,0-8), the higher the score, the more painful the patient feels
Sleep quality score the day transfer out of ICU | The day transfer out of ICU, an average of 1day
  Sleep quality score the day transfer out of ICU, assessed using St.Mary'sHospitalSleepQuestionnaire(SMHSQ, 11 to 55), the lower the score, the higher the degree of sleep disorders
Cognitive assessment score 60 days after surgery | Day 60 after surgery, an average of 1 day
  Cognitive assessment score 60 days after surgery, assessed using Telephone Interview for Cognitive Status-Modified(TICS-m,0-50), the higher the score, the better the cognitive function
Sleep quality score 60 days after surgery | Day 60 after surgery, an average of 1 day
  Sleep quality score 60 days after surgery, assessed using Pittsburgh sleep quality index(PSQI,0-21), the higher the score, the worse the sleep quality
ICU LOS | The day the patient transfer out of ICU, an average of 1 day
  ICU length of stay
Hospital LOS after surgery | The day the patient discharge, an average of 1 day
  Hospital length of stay after surgery
All cause mortality 60 days after surgery | Day 60 after surgery, an average of 1 day
  All cause mortality 60 days after surgery
Non-neurological complications 60 days after surgery | Day 60 after surgery, an average of 1 day
  Non-neurological complications 60 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jianxin Zhou, doctor, Study Chair — Beijing Shijitan Hospital, Capital Medical University
Locations (1):
- Beijing Shijitan Hospital.CMU, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No